CLINICAL TRIAL: NCT05916482
Title: Characterization of Vietnamese Patients With Obesity at Outpatient Clinics
Status: Completed | Type: Observational
Sponsor: University Medical Center Ho Chi Minh City (UMC) (Other)
Collaborators: Mỹ Đức Hospital (Other)
Responsible Party: Principal Investigator, Tran Quang Nam, Head of department of Endocrinology, University Medical Center Ho Chi Minh City (UMC)
Other Study IDs: WO/BVDHYD/1/23
Record Dates: First submitted 2023-05-12; First posted 2023-06-23 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Obesity
Keywords: Obesity; Vietnamese patients with obesity; Outpatient clinic
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OPT OBESE: Vietnamese patients with obesity present at outpatient clinics of University Medical Center Ho Chi Minh City and My Duc General Hospital

SUMMARY:
In the past three decades, obesity has emerged insurmountably, not only in affluent nations but also in many low- and middle-income countries worldwide. It has been linked to various non-communicable diseases, including hypertension, coronary heart disease, diabetes mellitus, dyslipidemia, stroke, colorectal cancer, and many other chronic conditions, such as musculoskeletal disorders, putting tremendous pressure on healthcare systems and the socio-economy. The Asia and Pacific region harbors the highest absolute number of people with overweight and obese, amounting to approximately 1 billion. In Southeast Asia, the prevalence of overweight and obesity increased by almost 40% between 1990 and 2013. Although Vietnam has the lowest percentage of obese adults in the region (about 3.6%), we experienced a 38% increase in the number of obese people between 2010-2014, much higher than that in the University Kingdom and the United States (10% and 8% correspondingly). However, the problem is underestimated by not only healthcare professionals but also patients with obesity. These alarms underscore the necessity of implementing a comprehensive assessment and more focused and practical strategies for addressing obesity in Vietnam, where data has been limited. Therefore, our research has two arms: (1) characterization of patients with obesity to identify those at the highest risks for obesity complications, and (2) understating the attitudes and perceptions of people living with obesity to gain insights into the psychological factors associated with obesity. This research will be a foundation for further research on obesity in Vietnam and Southeast Asia.

DETAILED DESCRIPTION:
All Vietnamese, aged 18-65, diagnosed with obesity defined by BMI ≥ 25 kg/m2 as per Asia-Pacific Guidelines for Obesity, present at University Medical Center Ho Chi Minh City and My Duc General Hospital outpatient clinics, will be enrolled to the study. The patients will have:

* Standard anthropometric data will be done, using a professional medical HM200P Portable Height Stadiometer and a standardised ISO (International Organization for Standardization) 9001:2015 weight scale, by professional and experienced physicians according to standard study protocol: Weight, height, waist and hip circumference, waist to hip ratio, BMI calculated, followed by World Health Organization guidelines for Asian people.
* Blood pressure measure.
* Fat mass measured by the Tanita MC-780 MA (Serial: 17050004).
* Blood tests: fasting plasma glucose, cholesterol, HDL-C, LDL-C, and triglyceride.
* Mood disorder screening by answering a Patient Health Questionnaire-9.

ELIGIBILITY:
Inclusion Criteria:

* Subject is diagnosed with obesity defined by BMI ≥ 25 kg/m2

Exclusion Criteria:

* Inability to cooperate with height measurement.
* Inability to answer questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Vietnamese, aged 18-65, diagnosed with obesity defined by BMI ≥ 25 kg/m2 as per Asia-Pacific Guidelines for Obesity, present at University Medical Center Ho Chi Minh City and My Duc General Hospital outpatient clinics will be enrolled to the study.
Sampling Method: Non-Probability Sample
Enrollment: 502 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Weight measurement | At baseline
  Using standardized weight scale (ISO 9001:2015)
Height measurement | At baseline
  Using a professional medical HM200P Portable Height Stadiometer
Body Mass Index | At baseline
  Weight in kilograms divided by height in meters squared
Waist circumference | At baseline
  To be measured at the approximate midpoint between the lower margin of the last palpable rib and the top of the iliac crest
Hip circumference | At baseline
  To be measured around the widest portion of the buttocks.
Blood pressure | At baseline
  Systolic and diastolic pressure measurements will be taken using a standardized sphygmomanometer.
Fasting plasma glucose | At baseline
  Fasting plasma glucose (mmol/L) concentrations in serum
HDL cholesterol | At baseline
  HDL cholesterol (mmol/L) concentrations in serum
LDL cholesterol | At baseline
  LDL cholesterol (mmol/L) concentrations in serum
Triglycerides | At baseline
  Triglycerides (mmol/L) concentrations in serum
Total cholesterol | At baseline
  Total cholesterol (mmol/L) concentrations in serum
Body composition change | At baseline
  Body fat mass (% BFM), body fat percentage (%BF), muscle mass, skeletal muscle mass (% SMM) and visceral fat rating will be evaluated to assess body composition change. Measurements will be assessed using a Electrical bioimpedance (BIA)
Risk of depression score | At baseline
  Risk of depression will be assessed using PHQ-9 (Patient Health Questionnaire-9). It is scored on a 27-point scale. Those with a PHQ-9 score less than five is considered at no risk of depression, and those with a PHQ-9 score equal to or more than 5 are at risk of depression.

SECONDARY OUTCOMES:
The relationship between the severity of obesity to anthropometric parameters | At baseline
  The correlation between the severity of obesity to anthropometric parameters (waist circumference, hip circumference, weight, height, and BMI) will be evaluated.
The relationship between the severity of obesity to biochemical parameters | At baseline
  The correlation between the severity of obesity to biochemical parameters (fasting plasma glucose, LDL cholesterol, HDL cholesterol, triglycerides, and total cholesterol) will be evaluated.
The relationship between the severity of obesity to body composition | At baseline
  The correlation between the severity of obesity to body composition (body fat mass (% BFM), body fat percentage (%BF), muscle mass, skeletal muscle mass (% SMM) and visceral fat rating) will be evaluated.
The relationship between the severity of obesity to risk of depression | At baseline
  The correlation between the severity of obesity to risk of depression (PHQ-9 score) will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Nam Q Tran, MD, PhD, Principal Investigator — University Medical Center Ho Chi Minh City (UMC)
Locations (2):
- Vietnam (2):
  - My Duc General Hospital, Ho Chi Minh City
  - University Medical Center Ho Chi Minh City (Umc), Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/82/NCT05916482/Prot_000.pdf
  • Informed Consent Form (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/82/NCT05916482/ICF_001.pdf